CLINICAL TRIAL: NCT05818696
Title: A Brief Fear of Uncertainty-Focused Intervention as an Adjunct to Lethal Means Counseling
Brief Title: Uncertainty and Firearms: Obtaining Secure Storage
Acronym: UFOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Rutgers University (Other)
Responsible Party: Principal Investigator, Nicholas Allan, Research Assistant Professor, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PR210299
Record Dates: First submitted 2023-03-02; First posted 2023-04-19 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: All participants receive both interventions but the order in which a participant receives the interventions is randomized.
Who Masked: Outcomes Assessor
Masking Description: Raters completing the outcome assessments will be blind to condition.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LMC - CUE (Experimental): In this arm, participants will receive Lethal Means Counseling before receiving CBT for Uncertainty-Enhanced (CUE).
  Interventions: Behavioral: Lethal Means Counseling (LMC); Behavioral: CBT for Uncertainty - Enhanced (CUE)
- CUE - LMC (Experimental): In this arm, participants will receive CBT for Uncertainty-Enhanced (CUE) before receiving Lethal Means Counseling.
  Interventions: Behavioral: Lethal Means Counseling (LMC); Behavioral: CBT for Uncertainty - Enhanced (CUE)

INTERVENTIONS:
Behavioral: Lethal Means Counseling (LMC) — The research interventionist uses a guiding approach to identify methods for secure firearm storage and reflects the participant's reasons for and against secure firearm storage, with a particular focus on the service member's verbalized reasons for wanting to adopt or use the identified storage methods.
Behavioral: CBT for Uncertainty - Enhanced (CUE) — CUE consists of a 1-hour manualized intervention that uses interactive content to enhance participant learning of critical intervention components. The session includes (1) psychoeducation regarding the role of IU in exacerbating anxiety/mood sensations, (2) practice identifying and challenging maladaptive thoughts about uncertainty and accompanying distress, and (3) behavioral activities to challenge participants' capacity to handle uncertainty.

SUMMARY:
The goal of this clinical trial is to test whether inclusion of cognitive behavioral therapy (CBT) for Uncertainty-Enhanced (CUE) with Lethal Means Counseling (LMC) is acceptable, feasible, and efficacious in addressing secure firearm storage and associated psychological constructs in active duty servicemembers. The clinical trial aims to:

* Assess the preliminary efficacy of a LMC intervention, augmented with CUE, on firearm storage practices
* Examine mechanisms through which CUE and LMC increase firearm storage practices
* Assess credibility and acceptability of LMC

Participants will complete:

* One baseline visit
* Two intervention sessions-CUE and LMC
* Six brief surveys per day for 28 days using a mobile application
* One mid-point survey and five follow-up surveys

DETAILED DESCRIPTION:
Firearms are the leading cause of death in US suicides and account for more than 60% of military suicides. A primary driver of these high rates appears to be ready access to firearms. Research suggests that firearm suicides could potentially be reduced by reducing and/or limiting access to firearms. Considering these data, lethal means counseling (LMC) is a recommended best practice for suicide prevention (e.g., National Action Alliance for Suicide Prevention). Results of a recently completed Department of Defense-sponsored randomized control trial (RCT) conducted by the investigators showed that safe firearm storage practices (i.e., use of locking devices and/or safes) could be increased among Servicemembers using a brief lethal means counseling (LMC) protocol developed in part by the investigators. Though superior to control, 45% of Servicemembers who received LMC still maintained at least one unsafely stored firearm, suggesting they continued to experience barriers to behavior change. Accumulating evidence suggests that fear of the unknown-a form of anxiety commonly experienced by people with low tolerance for uncertainty-may be an important barrier to safe firearm storage. The primary aim of Project 5 is to test a brief modular intervention to improve the effectiveness of LMC on safe firearm storage practices among firearm-owning Servicemembers. In this study, the investigators will examine if LMC's effects on firearm storage practices can be enhanced among Servicemembers who first receive an intervention designed to reduce their intolerance of uncertainty (IU). These results could provide important information about how LMC can be most effectively delivered to an especially high risk subgroup of firearm-owning Servicemembers.

F1.1. Firearm Acquisition and Storage as a Strategy to Cope with Fear of the Unknown. The coping model of protective gun ownership posits that people acquire firearms to reduce distress experienced from inflated perceptions of environmental threat, and are unlikely to safely store firearms because doing so is perceived to inhibit readiness to respond to unexpected and uncertain threats. Firearm owners who acquire firearms for the primary purpose of self-protection (i.e., protective firearm owners) report overgeneralized perceptions of the world and other people as dangerous and/or threatening. Among firearm owners, exaggerated threat perceptions are also associated with the intention to acquire additional firearms. Negative affect is significantly higher among firearm owners who use no safe storage practices (F(1,872)=6.9, p=.009). Anxiety about the unknown may therefore serve as a barrier to safe firearm storage and decrease the effectiveness of LMC. The investigators will test this hypothesis by testing the impact of a brief intervention designed to reduce IU when delivered to firearm-owning Servicemembers.

F1.2. Intolerance of Uncertainty as a Risk Factor for Anxiety and Unsafe Firearm Storage. IU involves an aversion to ambiguity and increased distress when experiencing uncertainty. Elevated IU amplifies the experience of stress and anxiety, causing people to engage in maladaptive cognitive and behavioral strategies to reduce distress. It is posited that IU may impact a Servicemember's perception of threat from the environment and that this heightened threat perception will limit their desire for safe storage practices. This is supported by a recent study by the investigators in which IU and exaggerated threat expectancy were significantly higher among adults intending to acquire a firearm as compared to those who were not (partial η2=.014-.017). Among Servicemembers with elevated IU, adoption of safe firearm storage practices may therefore be enhanced if IU is first reduced. This hypothesis will be tested in the current study using an empirically-supported, brief web-based intervention. The use of a web-based intervention platform significantly improves the potential scale and reach of the intervention.

F1.3. Targeting IU to Enhance Lethal Means Counseling (LMC). IU is an ideal construct to target in a web-based intervention given the abundance of research finding elevations in IU across a broad spectrum of suicide risk factors. For example, IU is a strong transdiagnostic correlate of many psychological and behavioral disorders associated with increased risk for suicide: generalized anxiety disorder, major depression, obsessive compulsive disorder, social anxiety disorder, panic disorder and agoraphobia, substance use disorders, eating disorders, and posttraumatic stress disorder. Other studies have implicated IU as a risk factor for suicidal thoughts and behaviors. IU is malleable, even in very brief interventions. In a recent study, the investigators conducted the only RCT of a CBT-based intervention for IU. In that study, an in-person IU Treatment (IUT) comprised of psychoeducation and cognitive reappraisal techniques was compared to a control condition focused on psychoeducation about health lifestyle behaviors. IUT led to significantly larger reductions in IU, anxiety, and depression during follow-up, indicating IU can be reduced with a brief intervention. Results of that study also showed that the majority of participants found the intervention easy to understand, helpful, and applicable to their daily lives.

F1.4. IUT Refinement. Since completing this first RCT, this intervention has been refined to improve the intervention. When modifying interventions, it is critical to involve relevant stakeholders in the process. Two key alterations to IUT include a web-based delivery and augmenting IUT with a mobile app for ecological momentary assessment (EMA) and ecological momentary intervention (EMI). EMI is ideal for these brief interventions because it allows for participants to gain much-needed practice of challenging negative automatic thoughts and completing behavioral experiments in real-time, thereby improving internalization of learned skills and strategies. The investigators recently completed a focus group with 8 people (M age = 33.13, standard deviation [SD] = 11.50; 62.5% female) reporting IU at least 1 SD above the community mean (M = 43.75, SD = 7.5). Participants reported the content was accessible, easily understood, and highly relevant to their distress. Participants thought inclusion of EMA and EMI would improve participant engagement and reported they would not perceive completion of multiple surveys daily to be a burden. Participants also believed that personalized content would increase engagement. Finally, participants assisted in identifying exemplar behavioral experiments and in refining a delivery mechanism as successful completion of behavioral experiments is a core driver in anxiety-based CBT interventions. Similar augmentations to brief interventions for stress (d = .5), generalized anxiety disorder (ds = .4-.6), and panic disorder (d = .5) have been successful in enhancing intervention effects, further underscoring the promise of including EMI to optimize outcomes.

F1.5. Summary. In a recently completed RCT, the investigators showed that LMC increases firearm storage practices among firearm-owning Servicemembers. Despite these promising results, nearly half of Servicemembers did not fully adopt safe firearm storage practices. Subsequent research suggests that exaggerated perceptions of the world as a dangerous and threatening place may be a barrier to these practices. This study is designed to determine if a brief intervention that has been shown to reduce IU-a cognitive bias that increases threat perceptions and anxiety-can increase the effectiveness of LMC. This project will be the first to test a brief modular intervention to improve LMC as a preventative intervention for suicide. These results could inform community-based suicide prevention efforts in the DoD and may also improve the effectiveness of LMC delivered within healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

* are currently serving in any Branch or Component of the U.S. military, or were discharged from the U.S. military within the past 90 days
* 18 years or older
* Intolerance of uncertainty scale-12 total score equal to or greater than 35 (i.e., one SD above the community mean)
* own at least one firearm located in their home or vehicle that is stored unlocked and loaded (i.e., not secure storage)
* are able to speak and understand the English language

Exclusion Criteria:

* do not pass the Informed Decision Making Capacity (IDMC) screener, suggesting severe cognitive impairment
* have a psychiatric or medical condition that would prevent them from providing informed consent or from participating in the treatments (e.g., psychosis, mania, acute intoxication)
* no or limited access to an Android or Apple smartphone that is compatible with the EMA application

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Researcher developed items capturing changes in firearm storage practices | Change will be assessed from baseline to a) two weeks after the first intervention (midpoint) (b) two weeks after the second intervention (postintervention) and (c) six months after the first intervention (6 month followup)
  Firearm storage practices are assessed by asking participants: How often are the following specific firearm storage practices used (1) stored using a locking device, (2) stored in a locked location (e.g., lockbox, gun safe), (3) stored loaded. Questions are rated from never (0%) to always (100%) with higher scores indicating greater percentage using particular firearm storage practices.

SECONDARY OUTCOMES:
Credibility/Expectancy Questionnaire | Four weeks after the first intervention session (postintervention)
  Satisfaction with the interventions is measured using the Credibility/Expectancy Questionnaire (CEQ). The CEQ measures credibility and expectancy with a 6-item measure. Each item is measured on a 9-point scale from 1 to 9 with higher scores indicating a more positive rating. Scores range from 6 to 54.
Patient Satisfaction Questionnaire | Four weeks after the first intervention session (postintervention)
  Satisfaction with the interventions is measured using the Patient Satisfaction Questionnaire (PSQ). The PSQ measures patient satisfaction using an 11-item measure. Each item is measured on a 5-point scale from (1) Strongly Disagree to (5) Strongly Agree. Higher scores indicate greater satisfaction with the intervention components with scores ranging from 11 to 55.
Change in Intolerance of Uncertainty-12 scale score | Change will be assessed from baseline to a) two weeks after the first intervention (midpoint) and two weeks after the second intervention (postintervention)
  Intolerance of uncertainty is measured using the 12-item Intolerance of Uncertainty Scale - Short Form. Each item is measured on a 5-point scale from (1) Not At All Characteristic Of Me to (5) Entirely Characteristic Of Me. Higher scores indicate worse intolerance of uncertainty with scores ranging from 12 to 60.
Change in Intolerance of Uncertainty - Implicit Bias | Change will be assessed from baseline to a) two weeks after the first intervention (midpoint) and two weeks after the second intervention (postintervention)
  Intolerance of uncertainty is measured using an Implicit Association Test (IAT-Intolerance of Uncertainty). The test includes 20 items across four stimuli categories. Implicit association test (IAT) scores were calculated according to the algorithm developed by Greenwald, Nosek, and Banaji (2003) to combine accuracy and RT (across practice and test trials) into a single value. Using this algorithm IAT-IU scores of zero indicate no bias, positive scores indicate a bias toward pairing self-words with IU-words, and negative scores indicate a bias toward pairing self-words with certain-words.
Change in Firearm Implicit Bias | Change will be assessed from baseline to a) two weeks after the first intervention (midpoint) and two weeks after the second intervention (postintervention)
  Bias towards firearms is measured using an Implicit Association Test (IAT-Firearms). The test includes 20 items across four stimuli categories. IAT scores were calculated according to the algorithm developed by Greenwald, Nosek, and Banaji (2003) to combine accuracy and RT (across practice and test trials) into a single value. Using this algorithm IAT scores of zero indicate no bias, positive scores indicate a positive bias regarding firearm storage practices, and negative scores indicate a negative bias regarding firearm storage practices.
Researcher developed questions assessing change in openness to utilize firearm storage practices | Change will be assessed from baseline to a) two weeks after the first intervention (midpoint) (b) two weeks after the second intervention (postintervention) and (c) six months after the first intervention (6 month followup)
  Openness to utilize firearm storage practices are assessed by asking participants: How open are you to engage in the following specific firearm storage practices (1) store using a locking device, (2) store in a locked location, (3) store unloaded. Questions are rated from not at all (1) to extremely open (5). Participants may also respond 'I already store all of my firearms in this manner.' Higher scores indicate a greater willingness to utilize certain firearm storage practices.

OTHER OUTCOMES:
Researcher developed questions assessing Firearm Acquisition | four weeks after the intervention and 3, 6, 9, and 12-month follow-up
  Researcher-developed items inquiring about firearm acquisition between assessment appointments. This is a count variable indicating the number of guns acquired.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University Department of Psychiatry and Behavioral Health, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified demographic and clinical data collected as part of this project will be available as raw individual-level data for sharing with external researchers working at an institution with a Federalwide Assurance (FWA) for the Protection of Human Subjects. Data will therefore be available for secondary analytic purposes. Names and institutions of persons either given or denied access to data will be tracked by our Administrative Core and will be available upon request from the sponsor. Data will not be available for data sharing until after this project is complete and the primary outcomes are published.
Supporting Information: Study Protocol
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for at least the next two years. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial individual participant data (IPD) can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).